CLINICAL TRIAL: NCT04853160
Title: Drug Utilization Study to Describe the Pattern of Febuxostat Use in Relationship to Allopurinol Following Addition of the Boxed Warning and Modification of the Indication Based on the Results of the CARES Trial
Brief Title: Drug Use Study of Febuxostat After Recent Changes in the Prescribing Information
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: Febuxostat-5006
Record Dates: First submitted 2021-04-20; First posted 2021-04-21 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Gout; Cardiovascular Diseases
MeSH Terms: conditions — Gout; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All Participants With Gout: Participants with gout, initiating febuxostat therapy on or after 01 June 2016 will be included in the study.

SUMMARY:
The prescribing information provides information on medicines. This study will check the number of patients starting febuxostat and the number of febuxostat users with cardiovascular disease after changes to the prescribing information.

DETAILED DESCRIPTION:
This is a descriptive, cross-sectional, non-interventional study of participants with gout. The study will evaluate the impact of the 2019 labeling changes (boxed warning and modified indication), based upon results of the cardiovascular safety of febuxostat and allopurinol in participants with gout and cardiovascular morbidities (CARES) trial, on febuxostat utilization.

The study will evaluate data from approximately 24046 participants. The data will be collected from optum clinformatics dataMart (CDM) including the medicare advantage administrative US claims database and the IQVIA pharmetrics plus claims database.

All participants will be enrolled in a single observational cohort. This trial will be conducted in the United States. The overall duration of this study is approximately 14 months.

ELIGIBILITY:
Inclusion Criteria:

1. Index fill date on or after 01 June 2016.
2. Having at least one diagnosis for gout (identified with diagnosis codes, International Classification of Diseases, clinical modification, ninth revision [ICD-9-CM]: 274.x or International Classification of Diseases, tenth revision [ICD-10]: M10.x) at any time in the participant's record.
3. Continuously enrolled for at least 12 months prior to index fill date.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with gout initiating febuxostat therapy on or after 01 June 2016 will be observed.
Sampling Method: Non-Probability Sample
Enrollment: 24046 (Actual)
Dates: Start 2020-08-15 (Actual); Primary Completion 2021-01-05 (Actual); Study Completion 2021-01-05 (Actual)

PRIMARY OUTCOMES:
Number of Participants Newly Initiating Febuxostat Therapy Versus Prevalent New Users | Up to 14 months
  Participants will be categorized into new users and prevalent new users. New users are participants who were naïve to allopurinol, defined as no record of allopurinol use in all historic pharmacy or medical claims at any time prior to initiation of febuxostat. Prevalent new users are participants who had used allopurinol and switched, defined as at least one record of allopurinol use in all historic pharmacy or medical claims at any time prior to initiation of febuxostat.
Number of Participants With Established Cardiovascular Disease (CVD) | Up to 14 months
  Participants initiating febuxostat will be categorized as having (Yes/No) to each of the following morbidities at any time prior to initiation of febuxostat: myocardial infarction (MI), unstable angina, stroke (hemorrhagic and ischemic), transient ischemic attack, peripheral vascular disease, diabetes mellitus with evidence of macrovascular or microvascular disease.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Central Contact, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/6082dfadf89629001e47b4db